CLINICAL TRIAL: NCT03651960
Title: Mobile and Interactive Robot's Social Acceptability for Balance and Gait
Brief Title: Mobile and Interactive Robot's Social Acceptability for Balance and Gait Rehabilitation
Acronym: ROBO-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 35RC12_9793; 2015-A00910-49 (Other: Id-RCB)
Record Dates: First submitted 2016-09-13; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Stroke Sequelae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot (Experimental): ROBOT PROTOTYPE
  Interventions: Other: ROBOT PROTOTYPE

INTERVENTIONS:
Other: ROBOT PROTOTYPE — The intervention consists of 12 45-minute sessions of balance and gait training with a mobile and interactive robot prototype for 4 weeks.

SUMMARY:
The recovery of a balance and gait is a primary objective for geriatric, neurological or orthopedic rehabilitation. Since the 80s, many walking robots were proposed.

Despite encouraging results, the use of robotic equipment for gait training remains limited, even if they meet a strong social demand. The reasons for this situation are economic, but also related to the non consideration of the context of utilization . It is therefore important to involve the users of the innovation in the development process because it is the latter that will broadcast. Psychosocial perspective of the acceptability of the technology meets this need by including the users' perceptions toward device (s).

The ROBO-K project aimed at developping a mobile and interactive robot, dedicated to the rehabilitation of balance and gait at an early stage. It was intended for patients with impaired walking vascular neurological, traumatic or associated with chronic neurological disease. The first step for its developement was conducted with the psychosocial approach of Technology acceptability which has required specific methods for collecting the views of users and analysis of the activity. This process allowed the design and the development of robot prototypes.

The aim of the present study is now to establish the degree of social acceptability of the robot and to analyze balance and gait training activity.

DETAILED DESCRIPTION:
The recovery of a balance and gait is a primary objective for geriatric, neurological or orthopedic rehabilitation. Since the 80s, many walking robots were proposed.

Despite encouraging results, the use of robotic equipment for gait training remains limited, even if they meet a strong social demand. The reasons for this situation are economic, but also related to the non consideration of the context of utilization (eg therapeutic practices , users' expectations). It is therefore important to involve the users of the innovation in the development process because it is the latter that will broadcast. Psychosocial perspective of the acceptability of the technology meets this need by including the users' perceptions toward device (s).

The ROBO-K project aimed at developping a mobile and interactive robot, dedicated to the rehabilitation of balance and gait at an early stage. It was intended for patients with impaired walking vascular neurological, traumatic or associated with chronic neurological disease. The first step for its developement was conducted with the psychosocial approach of Technology acceptability which has required specific methods for collecting the views of users and analysis of the activity. This process allowed the design and the development of robot prototypes. The aim of the present study is now to establish the degree of social acceptability of the robot and to analyze balance and gait training activity. The data collected will validate the development of assumptions with users (e.g. static or dynamic balance exercises, rehabilitation of gait in different paths).

The intervention consists of 12 45-minute sessions of balance and gait training with a mobile and interactive robot prototype for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS

  * Patients with neurologic acute or chronic disease responsible for gait or balance deficiency
  * Absence of important cognitive or mood disabilities
* PRACTITIONNERS Minimal 1 year of practice related to balance and gait training in a neurology department

Exclusion Criteria:

* PATIENTS Minors or patients older than 80 years, Weight more than 150 kg, Measuring less than 150 cm or more than190 cm, pregnant and lactating women, cognitive or major mood disorders Being unable to deliver their consent; Protected adults and persons deprived of liberty.
* PRACTITIONERS Having received information about the robot prototype prior to the study ; Have less than 1 year of practice related to balance and gait training in a neurology department; Protected adults and persons deprived of liberty.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Social acceptability of robot prototype for patient | Comparison of evaluations at baseline and up to 5 months
  This assessment is based on classical models of social acceptability (cf. references).
  It is carried out through semi-directive interviews with patients done before and atfer the use of the prototype (to study the acceptance process in the medium term).

SECONDARY OUTCOMES:
Social acceptability of robot prototype for practitioner | Comparison of evaluations at baseline and up to 5 months
  This assessment is based on classical models of social acceptability (cf. references).
  It is carried out through semi-directive interviews with practitioners done before and atfer the use of the prototype (to study the acceptance process in the medium term).
Evolution of the patient's self perception | Comparison of evaluations at baseline and up to 1 months
  Rosenberg self esteem scale : A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self.
  The scale is believed to be uni-dimensional. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BONAN, MD, PhD, Study Director — CHU Rennes
Locations (1):
- CHU de Rennes, Rennes, France

REFERENCES:
- [Background] Davis, F.D. (1989). Perceived usefulness, perceived ease of use, and user acceptance of information technology. MIS Quartely, 13 (3) : 319-340.
- [Background] Venkastesh, V., Morris, M.G., Davis, G.B. & Davis, F.D. (2003). User acceptance of information technology: toward a unified view. Mis Quartely, 27 (3), 425-478
- [Background] Heerink, M., Kröse, B., Evers, V., & Wielinga, B. (2010). Assessing acceptance of assistive social agent technology by older adults: the Almere Model. International Journal of Social Robotics, 2(4), 361-375
- [Background] Hamner, M. & Qazi, R. (2008). Expanding the technology acceptance model to examine personal computing technology utilization in government agencies in developing countries. Government Information Quaterly, 26(1), 128-136
- [Background] King, W.R., & He, J. (2006). A meta-analysis of the technology acceptance model. Information and Management, 43(6), 740-755
- [Background] Legris, P., Ingham, J., & Collerette, P. (2003). Why do people use information technology? A critical review of the technology acceptance model. Information and Management, 40(3), 191-204